CLINICAL TRIAL: NCT05518981
Title: The Clinical Significance of Patient Care Escalations From a Remote Monitoring Service
Brief Title: Effect of Remote Physiologic Monitoring (RPM) on Outcomes in COPD Patients
Status: Completed | Type: Observational
Sponsor: Spire, Inc. (Industry)
Collaborators: Pulmonary Associates of Richmond (Unknown); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: 20210406
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Acute Exacerbation of COPD; Hospitalization; Exacerbation; Remote Patient Monitoring; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Respiratory Remote Patient Monitor (Spire Health Tag) — The RPM service, tailored to chronic respiratory disease patients, utilizes a system that includes three components: undergarment-adhered cardiorespiratory sensors, in-home data transmission hub, and web-based clinical dashboard. The sensors are a set of six proprietary, skin-safe devices that include sensors for intermittent photoplethysmography, continuous respiratory force, and tri-axis accelerometers for activity. Clinical liaisons monitor deviations from patient-specific baselines and contact subjects for a "risk assessment" call, including questions about symptoms. If a subject fails the risk assessment, they are escalated to the site to be seen, and potentially treated, by their pulmonologist.

SUMMARY:
This pre/post study was a retrospective analysis of unplanned hospitalization rates in a cohort of COPD subjects started on remote physiologic monitoring (RPM) at a large, outpatient pulmonary practice. The study included all subjects with high healthcare utilization (≥1 hospitalization or emergency room visit in the prior year) who had elected to enroll in an RPM service for assistance with clinical management. Additional inclusion criteria included being on RPM for at least 12 months and a patient of the practice for at least two years (12 months pre- and post-initiation of RPM).

DETAILED DESCRIPTION:
This study included a retrospective analysis of data collected from subjects at a large outpatient pulmonology practice in the mid-Atlantic region of the United States between May 2019 and February 2022. At this clinic, patients who were candidates for RPM had been offered voluntary participation in service tailored to chronic respiratory disease patients (Spire Health, San Francisco, CA, USA). They continued regular follow-ups with their pulmonologists and received usual care according to the direction of their primary pulmonary physician for their COPD.

Inclusion criteria for the present study included a clinical diagnosis of COPD (COPD, chronic bronchitis, obstructive lung/airways disease, or emphysema), subscribed to RPM for at least 12 months as of February 28, 2022, full electronic medical records (EMR) at the site in question for one year before and one year after the start of RPM, and high healthcare utilization (≥1 ER visit or hospitalization in the year prior to enrollment). All such patients were included in the analysis.

The primary endpoint was unplanned, all-cause hospitalizations per subject. Secondary endpoints included unplanned cardiopulmonary hospitalizations, respective lengths of stay, ER visits, outpatient pulmonary visits, and systemic corticosteroid use, adherence to RPM, and time-to-visit (RPM escalation to provider visit).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD (COPD, chronic bronchitis, obstructive lung/airways disease, or emphysema)
* ≥1 hospitalization or emergency visit in the year prior to enrollment
* enrolled in the Spire RPM patient monitoring service for at least 12 months
* a patient of the practice for at least two years (12 months pre- and 12 months post-initiation of RPM).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COPD patients at a large outpatient pulmonology practice in the mid-Atlantic region of the United States. They were all candidates for RPM and were offered a voluntary participation in a service tailored to chronic respiratory disease patients.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
All-Cause Hospitalizations | 1 year pre- and 1 year post-initiation of RPM (2 years total)
  The change in number of all-cause hospitalizations per patient

SECONDARY OUTCOMES:
Cardiopulmonary Hospitalizations | 1 year pre- and 1 year post-initiation of RPM (2 years total)
  The change in number of cardiopulmonary hospitalizations per patient
All-Cause Emergency Room (ER) Visits | 1 year pre- and 1 year post-initiation of RPM (2 years total)
  The change in number of all-cause ER visits per patient
Cardiopulmonary Emergency Room (ER) Visits | 1 year pre- and 1 year post-initiation of RPM (2 years total)
  The change in number of cardiopulmonary ER visits per patient
Pulmonary Outpatient Visits | 1 year pre- and 1 year post-initiation of RPM (2 years total)
  The change in number of pulmonary outpatient visits per patient
Length of Stay | 1 year pre- and 1 year post-initiation of RPM (up to 2 years total)
  Length of hospitalization
Systemic Corticosteroid Use | 1 year pre- and 1 year post-initiation of RPM (2 years total)
  Number of new prescriptions of corticosteroids given by pulmonologist
Adherence to RPM | 1 year
  Proportion of days during the intervention period where physiological sensors were worn for at least 8 hours
Time to Visit | up to 1 year
  Time from escalation to visit with provider

CONTACTS AND LOCATIONS:
Overall Officials: Neema Moraveji, PhD, Principal Investigator — Spire Health
Locations (1):
- Spire, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided